CLINICAL TRIAL: NCT04010812
Title: The Effects of Discharge Readiness on Success Following Discharge From Sub-Acute Rehab
Brief Title: Effects of Discharge Readiness on Success Following Discharge From Sub-Acute Rehab
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Nancy Williams, Adjunct professor, Stony Brook University
Other Study IDs: 1352630-1
Record Dates: First submitted 2019-06-14; First posted 2019-07-08 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Discharge From Sub-acute Rehabilitation Facility
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — RHDS- Readiness For Hospital Discharge Scale, Patient Self-Assessment Form

SUMMARY:
Study's purpose is to determine if a patient's perception of readiness for discharge from sub-acute rehabilitation, as measured by Readiness For Hospital Discharge Scale Patient Self-Reports Form, correlates with the patient's success after discharge, measured by patient reported number of falls, emergency room visits and hospitalizations 30 days post discharge.

DETAILED DESCRIPTION:
All sub-acute rehabilitation patients will be approached for study participation one day prior to discharge day from the facility. Patients will be approached in their private room within the facility to obtain consent. Consent will be reviewed with patient by investigators. Patients will be asked to demonstrate understanding of the study and what consent will imply utilizing the teach back method. If patient is able to demonstrate understanding and gives consent the MoCA will be administered. If MoCA scores falls between 22-30 they will be included in study. If MoCA score falls below 22 they will not be included in study and that will be explained to them at that time. MoCA scores will be included in patient medical record. Patient name and assigned ID number, phone number, second contact and consent will be recorded on the confidential roster sheet and stored in a locked file cabinet located in director's office at Peconic Landing. The day of discharge patients will complete the RHDS survey. Investigators will complete the study data sheet including ID number, MoCA score, RHDS score, length of stay, discharge date, and recommended discharge therapy- home care, outpatient, none. Thirty to thirty-seven days after discharge investigators will call patient and ask 3 questions from scripted form. "How many falls have you had since discharge home:, "How many visits to the emergency room have you had since your discharge home","How many admissions to the hospital have you had since your discharge home." Following completion of telephone questions, confidential roster sheet and consent form will be shredded.

ELIGIBILITY:
Inclusion Criteria:

Montreal Cognitive Assessment score 22 or greater

* consent with observed teach back confirmation
* discharge from sub-acute rehabilitation

Exclusion Criteria:

* Montreal Cognitive Assessment score less than 22
* inability to "teach back" during consent process
* non english speaking

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Older adults discharged from a sub-acute rehabilitation facility
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2019-06-13 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of falls, ER visits, hospitalization | 30 days
  Participant reported 30 days after discharge from rehabilitation facility

CONTACTS AND LOCATIONS:
Locations (1):
- Peconic Landing, Greenport, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data Collection sheet